CLINICAL TRIAL: NCT03531463
Title: Nordic DeltaCon Trial: Non-operative Treatment Versus Reversed Total Shoulder Prosthesis in Patients Sixty Five Years of Age and Older With Displaced 3- and 4 Parts Proximal Humeral Fractures - a Prospective, Randomized Controlled Trial
Brief Title: The Nordic DeltaCon Trial for Displaced Proximal Humeral Fractures in Elderly
Acronym: DeltaCon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Tore Fjalestad, Principal investigator Tore Fjalestad, MD. Ph.D. Consultant Orthopaedic Surgeon, Mail: torfja@online.no / tofjal@ous-hf.no , Ph:+4797013389, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/476-D
Record Dates: First submitted 2018-04-27; First posted 2018-05-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Proximal Humeral Fracture
Keywords: Displaced; Non-Operative treatment; Reversed Total Shoulder Prosthesis
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blinded trial
Who Masked: Outcomes Assessor
Masking Description: Physiotheraphists specialized in shoulder injuries collect all data and perform all tests / interviews of patients during FU at 3 months, 1-2-5 years. Blinded for the allocation / treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative treatment (Active Comparator): Operative treatment of the displaced proximal humeral fracture with a reversed total shoulder prothesis (Delta prosthesis) using a stadardized deltopectoral approach, bone block grafting and thread cerclages of the tubercles.
  Rehabilitation with standardized physiotherapy guideline and self exercise protocol
  Interventions: Procedure: Operative treatment with Reversed Total Shoulder Prosthesis
- Non-Operative treatment (No Intervention): Rehabilitation with standardized physiotherapy guideline and self exercise protocol

INTERVENTIONS:
Procedure: Operative treatment with Reversed Total Shoulder Prosthesis — The standardized approach is the delto-pectoral to minimize any damage of the deltoid muscle. A cemented monoblock humeral stem will be implanted. Braided polyester suture-cerclages engaging the insertion of the subscapular and infraspinatus tendons enforced by a bonegraft or a "horseshoe-graft" from the humeral head will be used
  Arms: Operative treatment

SUMMARY:
The Nordic DeltaCon Trial is a prospective, single-blinded, randomized, controlled, multi-center and multi-national trial comparing reverse prosthesis and non-operative treatment in displaced proximal humerus fractures, in the elderly patients aged 65 to 85 years with displaced OTA/AO group B2 or C2 fractures (According to the new 2018 revision: AO/OTA (Orthopaedic Trauma Association) group 11-B1.1, 11-B1.2 and 11-C1.1, 11-C3.1. )

DETAILED DESCRIPTION:
Single-blinded, multi-center, multi-national (Finland, Sweden, Denmark, Norway) Primary outcome in this study is QuickDASH (The short form of Disabilities of the arm, shoulder and hand) score measured at two years.

Secondary outcomes are QuickDASH at/after one, two (short term) and five years (medium term), general visual analog scale (VAS) for pain, Oxford shoulder score (OSS), Constant-score (CS), number of re-operations and complications. Quality of life is assessed with 15-D. Cost-effectiveness analysis will be performed after completion of the trial.

In addition to 2 years main outcome (short term) follow-up will continue to 5 years (medium term) and 10 years (long term). The power calculation is based on 2 years.

ELIGIBILITY:
Inclusion Criteria:

Low energy AO/OTA group 11-B1.1, 11-B1.2 and 11-C1.1, 11-C3.1. Both B and C type includes subgroups: Displaced [2], Impacted [3] or Non impacted [4] from the universal modifiers list.

Exclusion Criteria:

Radiographic Mal-inclination Less than; varus 30°or valgus 45° Less than 50% contact between head fragment and meta-/diaphysis Head split fractures with more than 10% of the articular surface in the main head fragment.

Head split fractures (group 11-C3.2 and 11-C3.3) with more than 10% of the articular surface in the main head fragment.

Dislocation or fracture-dislocation of the gleno-humeral joint Pathological fracture

General

* Refuse to participate
* Age under 65 years of age, or over 85 years of age
* Serious poly-trauma or additional surgery
* Non-independent, drug/alcohol abuse or institutionalized (low co-operation)
* Contra-indications for surgery
* Does not understand written and spoken guidance in local languages
* Previous fracture with symptomatic sequelae in either shoulder
* Patients living outside the hospital's catchment area

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Quick-DASH | From enrollment to 5 years follow-up. Scale 1-4 points (Total point x answers given) x25. Lowest point best
  The short form of Disabilities of the arm, shoulder and hand

SECONDARY OUTCOMES:
Oxford Shoulder Score | From enrollment to 5 years follow-up. Scale 0 - 48, lowest score best.
  Shoulder specific patient self-assesment
15 D Quality of Life | From enrollemtn to 5 years follow-up. 15 questions, 5 levels, scale 0.000 - 1.000. Highest number best.
  15 Questions 5 levels Generic Score (Harri Sintonen)
Constant score (CS) | From enrollment to 5 years follow-up. Scale 0- 100 points. Highest best if only actual shoulder is scored..
  Functional outcome for the shoulder
VAS pain | From enrollement to 5 eyars follow-up. Scale 0-15 points, best equal zero points
  General visual analog scale (VAS) for pain
Radiographic + Computer Tomography scan (CT) | From enrollemnt to 5 years follow-up for plain radiographs. CT at enrollement and at 2 years.
  Plain radiographs 2 plane (true front + scapula Y view) and CT of injured shoulder
Patient involvement | 2 years
  The aim of the interviews will be to move towards patient-centered medicine by taking into account the goals, preferences and values of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ville Mattila, Professor, Study Chair — Professor in orthopedics and traumatology, Tampere University Chief of musculoskeletal department, Tampere University Hospital Visiting professor, Karolinska Institute, Stockholm
Locations (3):
- Aarhus University Hospital, Division of Orthopaedics, Aarhus, Denmark
- Tampere University Hospital, Division of Orthopaedics, Tampere, Finland
- Oslo University Hospital, Division of Orthopaedics, Oslo, Norway

REFERENCES:
- [Background] Launonen AP, Fjalestad T, Laitinen MK, Lahdeoja T, Ekholm C, Wagle T, Mattila VM; NITEP-group. Nordic Innovative Trials to Evaluate osteoPorotic Fractures (NITEP) Collaboration: The Nordic DeltaCon Trial protocol-non-operative treatment versus reversed total shoulder arthroplasty in patients 65 years of age and older with a displaced proximal humerus fracture: a prospective, randomised controlled trial. BMJ Open. 2019 Jan 29;9(1):e024916. doi: 10.1136/bmjopen-2018-024916. PMID 30700485
- See also: Trial website for patients, their relatives and health workers — https://oslo-universitetssykehus.no/avdelinger/ortopedisk-klinikk/ortopedisk-avdeling-ulleval/brudd-i-ovre-del-av-overarmsbeinet-proksimale-humerus-den-nordiske-deltacon-studien

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03531463/SAP_000.pdf